CLINICAL TRIAL: NCT04384068
Title: The Safety and Effectiveness of Tocilizumab in Rheumatoid Arthritis in Real-World Clinical Setting
Brief Title: The Safety and Effectiveness of Tocilizumab in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HS-1383
Record Dates: First submitted 2017-10-17; First posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-04

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; tocilizumab; safety
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chinese RA patients: Chinese RA patients who used tocilizumab in real world clinical practice

SUMMARY:
The aim of this study is to investigate the safety and effectiveness of tocilizumab (Actemra®) using Chinese Rheumatology Information Platform (CRIP) on Chinese Rheumatology Data Centre (CRDC, http://www.crdc.org.cn/) in Chinese RA patients.

DETAILED DESCRIPTION:
Tocilizumab (Actemra®) is a humanized monoclonal antibody targeting the human IL-6 receptor, which inhibits the binding of this cytokine to its receptor. It is the first monoclonal antibody developed for RA treatment with this mechanism of action and has been approved by regulatory authorities in China since 2013. Data from five phase III studies with over 4000 recruited patients have shown that tocilizumab at a dose of 8 mg/kg, in combination with methotrexate/DMARDs or as monotherapy, can produce a quick and clinically relevant improvement in RA signs and symptoms, health status, and prevent joint damage, for both patients who have not been previously treated with and refractory to methotrexate, other DMARDs or anti-TNF agents. However, in real-world clinical setting, the safety profile and treatment pattern with regard to the persistence on tocilizumab and the efficacy are not clear in China. The aim of this study is to investigate the safety and effectiveness of tocilizumab using Chinese Rheumatology Information Platform (CRIP) on Chinese Rheumatology Data Centre (CRDC, http://www.crdc.org.cn/) in Chinese RA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Patients with a diagnosis of RA according to the revised (2010) ACR criteria.
* Patients per treating physician's judgment to treat with Tocilizumab.
* Signed written informed consent

Exclusion Criteria:

* Patients are receiving or have received any investigational agent 4 weeks (or 5 half-lives of investigational agent, whichever is longer) prior to enrollment of this study.
* Subjects with contra-indications to Tocilizumab therapy as detailed in the label (with known hypersensitivity to Tocilizumab or accessories; or with active infections.).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 2500 participants will be enrolled in this study from Approximately 50 investigational centers in China. The study population will include patients with RA, according to 2010 ACR criteria, in whom the treating physician has made the decision to treat with Tocilizumab. Furthermore, patients must have given their informed consent and must not meet any of the exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2018-12-27 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoints change from baseline to week 52 | Baseline, Week 52
  Incidence of AEs, SAEs and AESIs with severity determined through use of NCI-CTCAE version 4.03 in full RA population, as well as the causalities between AEs and Tocilizumab.
Safety endpoints change from baseline to week 52 | Baseline, Week 52
  Incidence and severity of unexpected AE/ adverse drug reaction（ADR）in RA patients

SECONDARY OUTCOMES:
Proportion of RA patients achieving treatment target measured by DAS28, CDAI, SDAI. | Baseline, Week 52
  Effectiveness endpoints
Mean changes from baseline in Health Assessment Questionnaire Disability Index score | Baseline, Week 52
  Effectiveness endpoints ( It consists of 20 questions referring to 8 component sets. The questionnaire will be scored based on the instructions from the Stanford University Medical Center and higher scores mean a worse outcome).

OTHER OUTCOMES:
Proportion of patients still on TCZ treatment after treatment initiation. | Baseline, Week 52
  Exposure endpoints
Mean dose of tocilizumab | Baseline, Week 52
  Exposure endpoints
Mean duration (weeks) of tocilizumab treatment measured by the weeks of continuous tocilizumab administrated, regardless of dose reduction | Baseline, Week 52
  Exposure endpoints
Proportion of patients with dose decrease, dose discontinuation (subject stopped Tocilizumab treatment and did not take any administration of tocilizumab till the end of study) and dose interruption and the possible reason. | Baseline, Week 52
  Exposure endpoints
Mean dose interval as measured by weeks between tocilizumab infusions. | Baseline, Week 52
  Exposure endpoints
Proportion of patients discontinued from tocilizumab for safety and efficacy. | Baseline, Week 52
  Exposure endpoints

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China